CLINICAL TRIAL: NCT02545335
Title: Neutrophil Function During Combination Therapy With Protease Inhibitors in Chronic Hepatitis C
Brief Title: Neutrophil Function During Therapy With Protease Inhibitors in Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: HCV-neutrophil
Record Dates: First submitted 2015-07-29; First posted 2015-09-09 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to characterize neutrophil function in patients undergoing chronic hepatitis C triple therapy with protease inhibitors in comparison to dual therapy with peginterferon and ribavirin and with interferon free treatment regimen to thereby elucidate the possible mechanisms of protease-inhibitor associated infections.

DETAILED DESCRIPTION:
Chronic hepatitis C infection (CHC) is a major health problem, potentially leading to liver related mortality via complications of liver cirrhosis or hepatocellular carcinoma, and affects more than 185 million persons worldwide. Antiviral therapy evolved during the past 25 years from standard interferon, the combination with ribavirin and pegylated interferon (P/R) to the addition of protease inhibitors and is currently on the edge to an interferon-free era with the first such substances being approved in 2014. However, current standard therapy for CHC genotype 1 patients without cirrhosis consists of ribavirin and pegylated interferon (P/R) in combination with boceprevir (BOC) or telaprevir (TPV), which are direct acting antivirals and represent the first-generation protease inhibitors.

Triple therapy for CHC has been reported to be associated with a quantitative and qualitative increase in treatment-related (serious) adverse events compared to the former standard therapy without protease-inhibitors. Moreover, reports of serious infectious complications during triple therapy - especially in patients with acquired immune deficiencies like liver cirrhosis - that lead to considerable morbidity and mortality, have accumulated recently. The mechanisms of this increased susceptibility to infections remain unclear. However, BOC is known to inhibit neutrophil elastase activity.

Aims of this study were therefore to analyse infections that occurred in CHC outpatients during therapy in the study centre, to prospectively characterize neutrophil function in patients undergoing CHC triple therapy in comparison to dual therapy with peginterferon and ribavirin and to thereby elucidate the possible mechanisms of protease-inhibitor associated infections.

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C
* planned antiviral therapy

Exclusion Criteria:

* immunosuppressive medication
* active infection at baseline
* treatment with antibiotics within the last two weeks

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic hepatitis C undergoing antiviral therapy
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
neutrophil phagocytosis | 12 weeks
  phagocytosis of labelled E.coli

SECONDARY OUTCOMES:
number of infections | 12 weeks
  reported infections

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Statdlbauer, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

REFERENCES:
- [Result] Spindelboeck W, Horvath A, Tawdrous M, Schmerbock B, Zettel G, Posch A, Streit A, Jurse P, Lemesch S, Horn M, Wuensch G, Stiegler P, Stauber RE, Leber B, Stadlbauer V. Triple Therapy with First Generation Protease Inhibitors for Hepatitis C Markedly Impairs Function of Neutrophil Granulocytes. PLoS One. 2016 Mar 3;11(3):e0150299. doi: 10.1371/journal.pone.0150299. eCollection 2016. PMID 26938078
- [Result] Leber B, Balazs I, Horvath A, Posch A, Streit A, Spindelbock W, Feldbacher N, Stiegler P, Stauber RE, Rechberger GN, Kollroser M, Sattler W, Nusshold C, Stadlbauer V. Direct acting antiviral therapy rescues neutrophil dysfunction and reduces hemolysis in hepatitis C infection. Transl Res. 2021 Jun;232:103-114. doi: 10.1016/j.trsl.2020.12.005. Epub 2020 Dec 19. PMID 33352296